CLINICAL TRIAL: NCT03206892
Title: Laparoendoscopic Single-site Surgery Versus Conventional Multi-port Laparoscopy in Ovarian Drilling: A Randomized Controlled Trial
Brief Title: LESS Surgery Versus Conventional Multiport Laparoscopy in Ovarian Drilling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Bahaa Eldin Ahmed, assistant professor, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: LESS surgery AinShamsMH
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Successful Surgical Procedure; Operative Time; Cosmetic Outcome; Intra- and Post- Operative Complications
Keywords: LESS surgery; conventional multi-port laparoscopy; SILS; Single-site surgery; Covidien; laparoscopy; minimally invasive surgery; ovarian drilling; PCOS; Diagnostic laparoscopy

STUDY DESIGN:
Intervention Model Description: women fulfilled the inclusion criteria and consented will be included in the study and randomly assigned into two groups using computer random sequence generator.
Who Masked: Participant, Outcomes Assessor
Masking Description: using sequentially numbered, opaque sealed enveloped; each envelope contains the method of intervention according to the random sequence and will be opened just before the intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LESS surgery (Experimental): Laparoscopic ovarian drilling for polycystic ovary syndrome in infertile women using laparoendoscopic single-site surgery (single incision through the umbilicus using modified Hasson technique).
  Interventions: Device: laparoscopic ovarian drilling
- conventional multi-port laparoscopy (Active Comparator): laparoscopic ovarian drilling for polycystic ovary syndrome in infertile women using conventional multi-port laparoscopy (three port system using a closed technique on the umbilicus, left and right lower quadrant areas).
  Interventions: Device: laparoscopic ovarian drilling

INTERVENTIONS:
Device: laparoscopic ovarian drilling — laparoscopic ovarian drilling for polycystic ovary syndrome in infertile women comparing LESS surgery to conventional multiport laparoscopy

SUMMARY:
laparoendoscopic single-site surgery is compared to conventional multi-port laparoscopy for polycystic ovary syndrome in infertile women undergoing ovarian drilling as regards successful surgical procedure with less side effects

DETAILED DESCRIPTION:
Laparoendoscopic single-site surgery; one of the most recent advances in the field of minimally invasive surgery, is the use of a single incision in the umbilicus for laparoscopic surgeries, is compared to the conventional multi-port laparoscopy for polycystic ovary syndrome in infertile women undergoing ovarian drilling as regards successful surgical procedure without conversion to laparotomy or use of an additional port in the single site group. in addition to operative time, intra- and post- operative complications and cosmetic outcome.

ELIGIBILITY:
Inclusion Criteria:

* PCOS according to Rotterdam Criteria (2 out of 3):
* polycystic ovaries (12 or more follicles in each ovary and/or increased ovarian volume >10 cm3).
* oligo- or an-ovulation.
* clinical and/or biochemical hyperandrogenisim. After exclusion of other aetiologies for irregular cycles.
* Indications of laparoscopic ovarian drilling:
* clomiphene citrate- resistance or failure: failure to conceive after 6 to 9 cycles.
* other indications for laparoscopy.
* before gonadotropin administration to decrease risk of OHSS and multiple pregnancy.
* before ART to decrease risk of severe OHSS in women who previously had canceled IVF cycles due to OHSS risk or who suffered from OHSS in a previous treatment.

Exclusion Criteria:

* previous 2 or more laparotomies.
* chronic pelvic pain, endometriosis or pelvic inflammatory diseases to avoid pelvic adhesions and bias in the quantification of postoperative pain.
* High BMI (>35kg/m2)
* do not possess a native umbilicus.
* advanced gynaecological surgeries or malignant disorders (TLH, ALVH, laparoscopic myomectomy).
* contraindication to any laparoscopy like any medical condition worsened by pneumoperitoneum or Trendelnburg position.

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
successful surgical procedure | 1 hour (minutes)
  without conversion to laparotomy or the use of an additional port in the single-site group (number of ports).

SECONDARY OUTCOMES:
operative time | 1 hour (minutes)
  from trocar insertion to last skin stitch (minutes)
intraoperative blood loss | 24 hour after end of procedure
  amount of blood in the suction bottle (mL), drop in postoperative haemoglobin (g/dl)
intraoperative complications | 1 hour
  blood transfusion (number of units), bowel, bladder or ureteric injuries
postoperative hospital stay | 3 days
  number of days
postoperative pain | 1st day
  visual analogue scale (0-10 scale), number of postoperative analgesic ampules needed
postoperative complications | 1st week
  hematoma, wound infection, ileus, UTI
cosmetic outcome | day 1 and day 7
  scar image

CONTACTS AND LOCATIONS:
Overall Officials: Hesham M. Fathy, MD, Study Chair — Ain Shams University; Ahmed M. Bahaa Eldin, MD, Study Director — Ain Shams University; Haitham Fathy M., MD, Principal Investigator — Ain Shams University; Maya M. AbdelRazek, M. Sc., Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided